CLINICAL TRIAL: NCT05274386
Title: Evaluation of the Impact of SpO2 Averaging Time on Performance of an Automatic FiO2 Control System: a Randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Czech Technical University in Prague (Other)
Collaborators: Motol University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: PricoOptisatAvg
Record Dates: First submitted 2022-02-14; First posted 2022-03-10 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Neonatal Respiratory Distress; Very Low Birth Weight Infant
Keywords: SpO2 averaging time; pulse oximetry; automatic oxygen control
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Intervention Model Description: Subjects will be switched between 3 averaging times (4to6s-10s-16s) every 12 hours. The sequence will be assigned in random order. Each enrolled subject will continue in the study with regular changes in averaging time through the course of their need for A-FiO2.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Averaging time 4to6 s (Other): The SpO2 averaging time will be set to 4to6 s for the next 12 hours. All elements of care will be as routinely used, except the changing of the averaging time setting.
  Interventions: Device: Fabian ventilator with PRICO system (Acutronic Medical Systems AG, Hirzel, Switzerland); SpO2 averaging time set to 4to6 s
- Averaging time 10 s (Other): The SpO2 averaging time will be set to 10 s for the next 12 hours. All elements of care will be as routinely used, except the changing of the averaging time setting.
  Interventions: Device: Fabian ventilator with PRICO system (Acutronic Medical Systems AG, Hirzel, Switzerland); SpO2 averaging time set to 10 s
- Averaging time 16 s (Other): The SpO2 averaging time will be set to 16 s for the next 12 hours. All elements of care will be as routinely used, except the changing of the averaging time setting.
  Interventions: Device: Fabian ventilator with PRICO system (Acutronic Medical Systems AG, Hirzel, Switzerland); SpO2 averaging time set to 16 s

INTERVENTIONS:
Device: Fabian ventilator with PRICO system (Acutronic Medical Systems AG, Hirzel, Switzerland); SpO2 averaging time set to 4to6 s — The SpO2 averaging time will be set to 4to6 s for the next 12 hours.
  Arms: Averaging time 4to6 s
Device: Fabian ventilator with PRICO system (Acutronic Medical Systems AG, Hirzel, Switzerland); SpO2 averaging time set to 10 s — The SpO2 averaging time will be set to 10 s for the next 12 hours.
  Arms: Averaging time 10 s
Device: Fabian ventilator with PRICO system (Acutronic Medical Systems AG, Hirzel, Switzerland); SpO2 averaging time set to 16 s — The SpO2 averaging time will be set to 16 s for the next 12 hours.
  Arms: Averaging time 16 s

SUMMARY:
The aim of the study is to determine the preferred oximeter averaging setting during automated control of FiO2 (A-FiO2) in infants receiving respiratory support and supplemental oxygen.

DETAILED DESCRIPTION:
There are 7 different averaging time settings available with PRICO (Acutronic Medical Systems AG, Hirzel, Switzerland), but after over a year of experience there is no clear clinical impression of the best setting. Therefore, a small systematic study is needed to determine the optimal guidelines.

ELIGIBILITY:
Inclusion Criteria:

* All VLBW on respiratory support and oxygen requirements after 2 weeks of age in the NICU are eligible after parental informed consent is obtained.

Exclusion Criteria:

* Parental informed consent is not obtained
* Recording device for automated control of FiO2 is not available

Min Age: 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Percent time in SpO2 target range | 20 days of intervention on average
  Percent time in the intended SpO2 target range (compliance), at SpO2 <86% (safety), and at SpO2 >98% (safety).
  Period with SpO2 higher than the target range with FiO2 =0.21 will be included in the target range compliance and excluded from time above the target range.

SECONDARY OUTCOMES:
Effect of set SpO2 target range and mode of ventilation on the percent time in SpO2 target range, at SpO2 <86%, and at SpO2 >98%. | 20 days of intervention on average
  A general linear model will be used controlling for target range (based on gestational age), mode of ventilation (e.g. High-frequency oscillatory ventilation, Continuous mandatory ventilation, Continuous positive airway pressure, High-flow nasal cannula, and Nasal intermittent positive pressure ventilation), and subject.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Janota, PhD, Principal Investigator — Motol University Hospital; Thomas E Bachman, MSc, Principal Investigator — Czech Technical University in Prague; Veronika Rafl-Huttova, MSc, Principal Investigator — Czech Technical University in Prague; Jakub Rafl, PhD, Principal Investigator — Czech Technical University in Prague
Locations (1):
- Motol University Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available upon reasonable request